CLINICAL TRIAL: NCT05414812
Title: Intervening on Women's Health for Rural Young Breast Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Cancer Resource Center of the Desert (Unknown); El Centro Regional Medical Center (Unknown); Pioneers Memorial Healthcare District (Unknown)
Responsible Party: Principal Investigator, Hui-Chun Irene Su, Professor, University of California, San Diego
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: 800646; B27BB4247 (Other Grant/Funding Number: California Breast Cancer Research Program)
Record Dates: First submitted 2022-05-25; First posted 2022-06-10 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2024-11

CONDITIONS: Breast Cancer; Fertility; Contraception; Menopausal Symptoms
Keywords: Oncofertility
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Interrupted time series design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Multi-component oncofertility care intervention (Experimental): After the intervention implementation, all breast cancer patients presenting to oncology clinical visits that meet eligibility criteria will receive the multi-component oncofertility care intervention.
  Interventions: Behavioral: Multi-component oncofertility care intervention
- Usual Care (No Intervention): Prior to the intervention implementation, all breast cancer patients presenting to oncology clinical visits that meet eligibility criteria will receive usual care.

INTERVENTIONS:
Behavioral: Multi-component oncofertility care intervention — The intervention includes:
  1. Young breast cancer patients presenting to oncology visits will complete a clinic-based oncofertility needs screen with a member of the clinical team. This needs screen assesses i) desire to have a child in the future, ii) need for contraception, and iii) sexual health/menopause symptoms.
  2. A women's health survivorship care plan (SCP) in Spanish and English encompasses content on screening and management strategies for a) fertility concerns/pregnancy health; b) contraception; c) hot flashes and d) sexual health.
  3. Oncofertility navigation consists of one telehealth or in-person session with a social worker to: i) assess the patient's oncofertility needs, ii) review the women's health SCP, iii) provide support with the goal of engaging in oncofertility care.
  4. Oncofertility consultation as indicated via telehealth or in person will occur between the patient and reproductive specialist. Each consultation is estimated to be 1 hour.
  Arms: Multi-component oncofertility care intervention

SUMMARY:
The purpose of this study is to evaluate the effectiveness of a multi-component intervention to improve young breast cancer survivors' engagement in goal-concordant oncofertility care, concurrently with observing and gathering information on how the intervention is implemented. The investigators hypothesize that implementation of the intervention will result in increased young breast cancer survivors' engagement in goal-concordant oncofertility care.

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer (Stages 0-IV) diagnosis
* Primary language English or Spanish
* Receiving oncology care at participating clinical sites
* Living in Imperial County, California

Exclusion Criteria:

- Women who are pregnant at recruitment

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 81 (Actual)
Dates: Start 2021-10-15 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Medical record review of engagement in goal-concordant oncofertility care | 12 weeks after oncology visit
  Study staff will be trained to abstract the primary outcome of engagement in goal-concordant oncofertility care from the patient's medical records using standardized case report forms. Engagement in goal-concordant oncofertility care will be assigned to young breast cancer survivors who undergo: 1) oncofertility needs screen, complete a navigation session, receive the women's health survivorship care plan (SCP), and thereafter have no oncofertility needs; OR 2) oncofertility needs screen, complete a navigation session, receive the SCP, have an oncofertility need, undergo telehealth oncofertility consultation, and thereafter have no oncofertility services needs; OR 3) oncofertility needs screen, complete a navigation session, receive the SCP, have an oncofertility need, undergo telehealth oncofertility consultation, have an oncofertility services need, and thereafter uptake appropriate services.

CONTACTS AND LOCATIONS:
Overall Officials: H. Irene Su, MD, MSCE, Principal Investigator — University of California, San Diego
Locations (4):
- United States (4):
  - Pioneers Medical Health District, Brawley, California
  - Cancer Resource Center of the Desert, El Centro, California
  - El Centro Regional Medical Center, El Centro, California
  - University of California San Diego, La Jolla, California

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual participant data generated during the study will be available from the principal investigator (H. Irene Su) upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication.
Access Criteria: Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to the principal investigator (H. Irene Su).

REFERENCES:
- [Derived] Romero SAD, Palomino H, Ahmed SH, Peacher D, Urias A, Ramirez L, Yocupicio J, Gutierrez P, Flores Ortega RE, Reyes B, Kaiser BN, Hoyt H, Su HI. Intervening on women's health for rural young breast cancer survivors: A study protocol. Contemp Clin Trials. 2023 Jul;130:107215. doi: 10.1016/j.cct.2023.107215. Epub 2023 May 8. PMID 37164298